CLINICAL TRIAL: NCT01691612
Title: Role of the Isomerase Pin-1 in the Development and Treatment of Asthma
Acronym: Pin1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elliot Israel, MD, Physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012P001029
Record Dates: First submitted 2012-09-07; First posted 2012-09-25 (Estimated); Results first posted 2017-07-03 (Actual); Last update posted 2017-07-03 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: Role of Pin-1 enzyme in Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- D. pteronyssinus allergens (Experimental): Single arm study exploring the role of Pin-1 enzyme in development of Asthma. Bronchoscopy before and 48 hours after installation of D. pteronyssinus allergens into the lung segments
  Interventions: Biological: installation of D. pteronyssinus allergens

INTERVENTIONS:
Biological: installation of D. pteronyssinus allergens — We will perform bronchoscopy and segmental allergen challenges. Subjects will undergo bronchoscopy with segmental installation of 5 ml of D. pteronyssinus (DerP). BAL and lung biopsy of the allergen-challenged segments will be performed 48 hr later
  Other Names: D. pteronyssinus allergens exposure

SUMMARY:
Pin1 is activated in asthmatic airways, increasing cytokine mRNA stability and eosinophil survival. This study is designed to test whether the Pin1 enzyme regulates TLR/IL-1R signal pathways in multiple cells in asthma.

DETAILED DESCRIPTION:
The investigators will test their hypothesis that Pin1 regulates TLR/IL-1R signaling pathways in asthma by examining Pin1 and related pathway activation in BAL-derived eosinophils after house dust mite allergen challenge. The investigators will perform segmental allergen challenge. BAL and lung biopsy of the allergen-challenged segments will be performed 48 hr later and activation of Pin1 and related pathways will be examined.

ELIGIBILITY:
Inclusion criteria:

* Subjects 18-55 years of age, diagnosed with asthma for at least 1 year;
* And FEV1 > 70% predicted on only short acting beta agonists e.g albuterol
* And methacholine PC20 < 8 mg/ml
* Positive skin prick test to Dermatophagoides pteronyssinus(DerP)
* No prior history of intubation for asthma
* No use of inhaled corticosteroids for 1 month prior to entry

Exclusion criteria:

* Current smoking or smoking history of greater than 10 pack-years
* Any other clinically important comorbidity determined by the principal investigator to affect subject safety, including uncontrolled diabetes, uncontrolled coronary artery disease, acute or chronic renal failure, and uncontrolled hypertension that would increase the risk of significant adverse events during bronchoscopy,
* Worsening of asthma symptoms requiring treatment with steroids within 4 weeks of screening
* Respiratory infection within four weeks
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant or who are currently pregnant or lactating.

Unless they:

* Are women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner
* Are women whose partners have been sterilized by vasectomy or other means
* Use one acceptable birth control method. Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.
* Pre-existing lung disease other than asthma
* History of coagulation disorders or abnormal PT/PTT testing at screening
* History of immunodeficiency diseases, including HIV
* A disability that may prevent the patient from completing all study requirements
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Diagnosis of Hepatitis B or C.
* History of alcohol abuse (as determined by the principal investigator) within 6 months of screening.
* History of illicit drug abuse (as determined by the principal investigator) within 6 months of screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kun P Lu, M.D., PhD, Principal Investigator — Beth Israel Deaconess Medical Center; Elliot Israel, M.D, Principal Investigator — Brigham and Womens Hospital
Locations (1):
- Asthma Research Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | D. Pteronyssinus Allergens
Started | 14
First Visit (Allergen Challenge) | 8
Second Visit (Bronchoscopy) | 7
Completed | 7
Not Completed | 7
Not completed — deemed ineligible after 1st visit | 6
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | D. Pteronyssinus Allergens
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Percentage of Total White Blood Cell That Were Eosinophils at 48 Hours
Description: Measure Pin1 activity in BAL-derived eosinophils after House Dust Mite (HDM) allergen challenge:
  Eosinophils post-challenge change from pre-challenge is reported: absolute change = [eosinophils post (%) - eosinophils pre (%)]
Time Frame: from baseline to 48 hours
Measure: Median (Full Range); unit: percent of white blood cells
Arm/Group | D. Pteronyssinus Allergens
Number analyzed (Participants) | 7
percent of white blood cells | 82.11 [0.24 to 88.51]

2. Secondary Outcome: Percent Change From Baseline in the Percentage of Total White Blood Cell That Were Lymphocytes at 48 Hours
Description: Percent change in percentage of total white blood cell that were lymphocytes is measured from pre-challenge to post-challenge as: [100% * ((Post-Pre)/Pre)]
Time Frame: from baseline to 48 hours
Measure: Median (Full Range); unit: percent change
Arm/Group | D. Pteronyssinus Allergens
Number analyzed (Participants) | 7
percent change | -64.3 [-100 to 50]

3. Secondary Outcome: Percent Change From Baseline in the Percentage of Total White Blood Cell That Were Macrophages at 48 Hours
Description: Percent change in percentage of total white blood cell that were macrophages is measured from pre-challenge to post-challenge as: [100% * ((Post-Pre)/Pre)]
Time Frame: from baseline to 48 hours
Measure: Mean (Full Range); unit: percent change
Arm/Group | D. Pteronyssinus Allergens
Number analyzed (Participants) | 7
percent change | -82.4 [-89.3 to -5.9]

4. Secondary Outcome: Change From Baseline in the Percentage of Total White Blood Cell That Were Neutrophils at 48 Hours
Description: Neutrophils have some zero values pre-challenge, so absolute change is reported instead of percent change: post-pre from baseline to 48 hours
Time Frame: from baseline to 48 hours
Measure: Mean (Full Range); unit: percent of white blood cells
Arm/Group | D. Pteronyssinus Allergens
Number analyzed (Participants) | 7
percent of white blood cells | 3 [-5 to 19]

ADVERSE EVENTS:
Arm/Group | D. Pteronyssinus Allergens
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 6/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D. Pteronyssinus Allergens (N=14)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (2)
Headache (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
increased asthma symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes